CLINICAL TRIAL: NCT06247813
Title: Pilot Study: Impact of Biomarker-Guided Dietary Supplementation on Quality-of-Life Measures in Subjects With Chronic Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ethos Research & Development (Industry)
Responsible Party: Principal Investigator, Joshua Gunn, Chief Science Officer, Ethos Research & Development
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-02-637-1557
Record Dates: First submitted 2024-01-12; First posted 2024-02-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nerve Health (Experimental)
  Interventions: Dietary Supplement: Nerve Health Formula
- Oxidative Stress (Experimental)
  Interventions: Dietary Supplement: Redox Support Formula
- Inflammation (Experimental)
  Interventions: Dietary Supplement: Inflammation Support Formula

INTERVENTIONS:
Dietary Supplement: Inflammation Support Formula — Turmeric Extract (400mg), Bioperine (Black pepper, 10mg), Ashwagandha (500mg), and Olive Leaf Extract (250mg).
  Arms: Inflammation
Dietary Supplement: Nerve Health Formula — Hydroxocobalamin (Vitamin B12, 1000mcg), Pyridoxal-5-Phosphate (Vitamin B6, 50mg), LMethylfolate (400mcg) and Trimethyl Glycine (Betaine, 750mg).
  Arms: Nerve Health
Dietary Supplement: Redox Support Formula — N-Acetyl-L-Cysteine (500mg), CoQ10 (250mg), Acetyl-L-Carnitine (200mg), Alpha Lipoic Acid (200mg), Benfotiamine (300mg), Selenium (250mcg), Riboflavin (50mg), Zinc (15mg) and Copper (1.8mg).
  Arms: Oxidative Stress

SUMMARY:
The goal of this study is to use pain-specific urine biomarkers to evaluate how daily nutritional supplementation with biomarker guided formulas effect, quality of life and urinary biomarker scores in chronic pain patients. Assessing the effect of biomarker guided supplementation on pain specific biomarkers through changes in urinary biomarker scores may solidify the necessity for identifying deficiencies to create an individualized treatment plan for pain patients. This study aims to evaluate the effect of biomarker-guided supplementation on the three categories of urinary biomarkers using targeted ingredients specifically designed for oxidative stress, inflammation, and nerve health. This study provides subjects with one of three nutritional supplement formulas based on their specific urinary biomarker test results and assesses changes in their urinary biomarker levels and their quality of life as it relates to their pain over a 3-month period.

ELIGIBILITY:
Inclusion Criteria:

* Previously submitted a urinary biomarker sample and agreed to be contacted for research.
* Be seeking treatment for chronic pain as defined as symptoms persisting for ≥ 3 months.
* Be able to take oral medication and/or be willing to adhere to the supplement regimen.

Exclusion Criteria:

* Diagnosis of bacterial or viral infection during or 3 months prior to the study.
* Severe or untreated psychiatric disturbance and/or any psychiatric disorder that required hospitalization in the year prior to the screening visit.
* A history of cancer within 5 years prior to screening visit.
* Be pregnant or breast-feeding or have plans to become pregnant at any time during the study
* Participant has a known sensitivity or allergy to any of the ingredients in the study products.
* Participant has any dietary restriction that prevents the participant from consuming any of the ingredients in the study products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative urine biomarker levels. | 1 and 3 months of supplementation.
  Quantitative urine biomarker levels after 1 and 3 months of supplementation.
Quality-of-life measures. | 1 month of supplementation, 3 months and at 3 month follow up.
  Summary scores of quality-of-life measures, patient reported outcome measurement information system 29 (PROMIS-29); assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. For overall scoring of the test (i.e., adding each response) a higher score equals more of the concept being measured (e.g., more Fatigue, more Physical Function), meaning a worse outcome.
Quality-of-life measures. | 1 month of supplementation, 3 months and at 3 month follow up.
  Summary scores of quality-of-life measures, Short Form- 36 (SF-36); The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Coding of each item varies across the measure however all items are scored so that a high score defines a more favorable health state.

SECONDARY OUTCOMES:
Visual Analog Scale pain scores | 1 month, 2 months, 3 months and at 3 month follow up.
  Visual Analog Scale (VAS) pain scores are asked with 4 questions, current pain, worst pain, least pain and average pain since the subjects last visit. The scale is 0 to 10 where 0 is "no pain" and 10 is "worst imaginable pain", 10 would indicate a worse outcome.
Depression symptoms. | 1 month, 2 months, 3 months and at 3 month follow up.
  Percentage of subjects with a decrease in depression symptoms.
Anxiety symptoms. | 1 month, 2 months, 3 months and at 3 month follow up.
  Percentage of subjects with a decrease in anxiety symptoms.
Sleep quality score | 1 month, 2 months, 3 months and at 3 month follow up.
  Sleep quality (Pittsburg Sleep Quality Index (PSQI)) score (and subscale scores). The PSQI is a 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations.17 The 19 items are grouped into 7 components, including (1) sleep duration, (2) sleep disturbance, (3) sleep latency, (4) daytime dysfunction due to sleepiness, (5) sleep efficiency, (6) overall sleep quality, and (7) sleep medication use. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Profile of Mood States | 1 month, 2 months, 3 months and at 3 month follow up.
  Profile of Mood States (POMS) score (and subscale scores). The POMS is a 40 item questionnaire assessing mood. The scale is a 5 point scale ranging from "Not at All" (0), "A Little" (1), "Moderately" (2), or "Quite a Lot" (3) or "Extremely" (4). Scores for the seven subscales are calculated by summing the numerical ratings for items that contribute to each subscale. Two of the items on the Esteem-related Affect (ERA) subscale are reverse-scored prior to being combined with the other items. They are all added or subtracted based on the subscale (TMD = [TEN+DEP+ANG+FAT+CON] - [VIG+ERA]. ) to obtain total mood disturbance. A higher score would indicate a negative outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Gunn, PhD, Principal Investigator — Ethos Research and Development
Locations (1):
- Ethos Research and Development, Newport, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT06247813/ICF_001.pdf